CLINICAL TRIAL: NCT04025411
Title: Effectiveness of Computerized Device New of Visual Motor Simulation Versus Mirror Therapy in Hemiplegic Patients. SI-VIM Study
Brief Title: Effectiveness of Computerized Device New of Visual Motor Simulation Versus Mirror Therapy in Hemiplegic Patients.
Acronym: SI-VIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Saint-Etienne Métropole (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18CH200; 2019-A00041-56 (Other: ANSM)
Record Dates: First submitted 2019-07-17; First posted 2019-07-18 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: Stroke; Upper limb rehabilitation; Computerized mirror therapy; Hemiparetic; Mirror therapy
MeSH Terms: conditions — Stroke | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patient with stroke ischemic or hemorrhagic will be included. They will have visual motor simulation with the Intensive Visual Simulation 3 (IVS3) device and electroencephalography (EEG).
  Interventions: Device: Intensive Visual Simulation 3 (IVS3) device; Device: Electroencephalography (EEG)
- Control group (Active Comparator): Patient with stroke ischemic or hemorrhagic will be included. They will have simulation with the traditional Mirror Therapy (TM) and electroencephalography (EEG).
  Interventions: Device: traditional Mirror Therapy (TM); Device: Electroencephalography (EEG)

INTERVENTIONS:
Device: Intensive Visual Simulation 3 (IVS3) device — Visual motor simulation with the Intensive Visual Simulation 3 (IVS3) device will be realized and consist of 5 sessions per week for 4 weeks (20 minutes).
  The patient looks on a screen in front of him, mirroring the movements made by his healthy hand, while attempting to perform the same movement with his paretic hand.
  Other Names: Computerized Mirror Therapy (TM) device
  Arms: Experimental group
Device: traditional Mirror Therapy (TM) — Simulation with the traditional Mirror Therapy (TM) will be realized and consist of 5 sessions per week for 4 weeks (20 minutes).
  Arms: Control group
Device: Electroencephalography (EEG) — Electroencephalography (EEG) will be performed during the 1st, 6th, 11th, 16th and 20th session of their programme will be made in order to evaluate brain activity.

SUMMARY:
Mirror Therapy (TM) has been shown to be effective in motor rehabilitation of the hemiplegic upper limb, but its implementation in current clinical practice has several difficulties, both from the patient and physiotherapist point of view.

A new computerized Mirror Therapy (TM) device (Intensive Visual Simulation 3 (IVS3), Dessintey) which aims to solve the TM compliance problems and make it more efficient have been developed.

DETAILED DESCRIPTION:
The aim of this study is to compare the observance and efficiency of the Intensive Visual Simulation 3 (IVS3) therapy as compared to traditional Mirror Therapy (TM) in a population of hemiplegic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* First ischemic or hemorrhagic stroke for less than one year
* Not having reoffend
* Responsible for an initially complete hemiplegia,
* Upper-limb deficiency with the modified Frenchay Score below 70,
* Not neurological history other than stroke,
* Having signed the written consent
* Affiliated or entitled to a social security scheme

Exclusion Criteria:

* Patient who have not Magnetic Resonance Images (MRI) of the brain during stroke
* Having complete lesion of the primary motor cortex
* With an addiction to alcohol or drugs
* With psychiatric illness, cognitive impairment, uncontrolled disease / epilepsy, malignancy, severe renal or pulmonary impairment
* History of associated disabling general disease
* With associated cerebellar syndrome
* With clinical involvement of the brainstem
* Pregnancy in progress
* Patients under the protection of justice.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline Fugl-Meyer motor assessment score at 18 days, at 32 days, and at 60 days | Day: 0, 18, 32, 60
  Measured by Fugl-Meyer motor assessment score at baseline, at 18 days, at 32 days, and at 60 days.
  Fugl-Meyer score assesses the analytical motor skills of the upper limb with minimum score at 0 (hemiplegia) and maximum score at 66 (normal motor performance).

SECONDARY OUTCOMES:
Change from baseline modified Frenchay Arm Test score at 18 days, at 32 days, and at 60 days. | Day: 0, 18, 32, 60
  Measured by Frenchay Arm Test score at baseline, at 18 days, at 32 days, and at 60 days.
  Frenchay Arm Test score assesses functional improvement of the activities of the upper limb paretics with minimum score at 0 (total dependence) and maximum score at 100 (complete autonomy).
Change from baseline Barthel index at 18 days, at 32 days, and at 60 days. | Day: 0, 18, 32, 60
  Measured by Barthel index at baseline, at 18 days, at 32 days, and at 60 days. Barthel index assesses autonomy with minimum score at 0 (total dependence) and maximum score at 100 (complete autonomy).
Change from baseline Abilhand questionnaire at 18 days, at 32 days, and at 60 days. | Day: 0, 18, 32, 60
  Measured by Abilhand questionnaire at baseline, at 18 days, at 32 days, and at 60 days.
  Abilhand questionnaire will allow self-evaluation of the function of the upper limb in daily life with minimum score at 0 (difficulties in daily life) and maximum score at 46 (no difficulties in daily life).
Analysis of brain activity | Month: 2
  Measured by Electroencephalography (EEG) results.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal GIRAUX, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No